CLINICAL TRIAL: NCT04267107
Title: Managing Fatigue: The Individual Program in People Living With Parkinson's Disease- A Protocol for a Feasibility Study
Brief Title: Managing Fatigue in People With Parkinson's Disease
Acronym: MFIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Responsible Party: Principal Investigator, Tanya Packer, Dr.Tanya Packer, Professor, School of Occupational Therapy, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019-4954
Record Dates: First submitted 2020-02-06; First posted 2020-02-12 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease
Keywords: Parkinsons disease; Self-management; Fatigue management; Occupational therapy
MeSH Terms: conditions — Parkinson Disease | interventions — Conservation of Energy Resources; Self-Management; Occupational Therapy

STUDY DESIGN:
Intervention Model Description: This feasibility study will use a mixed-methods approach, nested in a pilot 2-arm randomized control design (experimental and no intervention control). We will collect qualitative and quantitative data simultaneously which will expand our understanding of the feasibility of the program.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants cannot be masked to study groups in this study. The researcher who is responsible for data collection and data analysis will be masked to group allocation.
  A research assistant will assign ID codes to each participant, manage the key to the ID codes. Feasibility questionnaire, only for experimental group, will be coded with participant ID codes.
  Participants will be instructed not to share any information on group allocation with the researcher during the assessments. Masking of the assessor will be monitored by reports of the assessor receiving any information during the assessments on the allocation of the participant. If there are multiple occurrences of this, a sensitivity analysis will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Managing Fatigue:The Individual Program (Experimental): Participants in the experimental group will receive the 6-week MFIP. Individuals in experimental group :
  * will participate in six one-to-one sessions (each takes 60 to 90 minutes)
  * will complete the Feasibility Questionnaire #1, after each session (10 questions) (Appendix 6)
  * will complete Feasibility Questionnaire #2 after completing all six-sessions (12 questions) (Appendix 7)
  * will complete the post-test measurement after completion of the program (approximately 60 minutes to complete)
  * will complete the follow-up measurement, three months after the completion of the program (approximately 60 minutes to complete)
  * will be advised to continue with their current healthcare services.
  * may participate in one focus group (one-hour session)
  Interventions: Other: Individual Managing Fatigue Program
- Control Group (No Intervention): Participants in the control group will not receive the IMFP and they will be advised to continue with their current healthcare services.
  Participants in the control group:
  * will complete post-test measurements after 6 weeks (approximately 60 minutes),
  * will complete the follow-up measurements three months later after completing the program (approximately 60 minutes).
  * will be advised to continue with their current healthcare services.
  Following the study, participants in the control group will be offered the manual of the program and a three-hour training workshop after (three months after the baseline testing). In this workshop, they will learn about the about the program, including the pre-session activities, in-session activities, and homework. This workshop will be conducted by occupational therapists.

INTERVENTIONS:
Other: Individual Managing Fatigue Program — The Individual Managing Fatigue Program includes six weekly sessions that focus on sleep, communication and body mechanics, activity stations, priorities and standards, and balancing daily schedule. Each session includes three parts: 1) a pre-session activity 2) in-session activities/information and 3) homework. Prior to coming to each session, participants will be asked to complete activities that will help them prepare for the in-session discussions. During each session participants will discuss and practice the topics most important to them. Based on their discussions, participants and therapists will decide on activities to complete during each session and as homework. The therapist will help the participant begin the homework at the end of each session, and the participant will finish it outside of the session at home. At the beginning of the following session, the therapist and participant will review the homework.
  Other Names: Energy conservation; Self-management; Occupational therapy
  Arms: Managing Fatigue:The Individual Program

SUMMARY:
This pilot study aims to evaluate the feasibility of Managing Fatigue: The Individual Program (MFIP) in people living with Parkinson's disease. The Managing Fatigue Program, a six-week, self-management energy conservation course, focuses on strategies that help people with fatigue to make changes to save and use their energy to accomplish their daily activities. Several studies have adapted and evaluated different delivery formats of the program in conditions similar to Parkinson's disease, demonstrating that the Managing Fatigue Program is effective in reducing fatigue impact, depression, sleep problems, and improving quality of life, participation and self-efficacy. While this program has been tested in people living with many chronic conditions there has been only limited inclusion of people living with PD. This feasibility study, using a mixed-methods approach, nested in a pilot randomized control design, will evaluate the feasibility of the Individual Managing Fatigue Program from the perspectives of people with Parkinson's disease, and prepare for a full-scale randomized controlled trial (RCT).

In this study, Managing Fatigue: The Individual Program (MFIP) will be delivered using videoconferencing. This feasibility study will use a mixed-methods approach, nested in a pilot two-armed randomized controlled design. Using a concurrent mixed-method design, we will collect two types of data (qualitative and quantitative) simultaneously, expanding our understanding of the feasibility of the program. Data will be collected using feasibility questionnaires developed by the research team, standard outcome measures, and group discussions. Multiple recruitment strategies will be used to recruit a convenience sample of 50 participants (25 in each group) from across the province of Nova Scotia, Canada. Eligible participants will be randomly assigned to either the control or experimental group using sealed envelopes. The study outcome measures will be administered three times during the study; pre-test, post-test after 6 weeks, and at three-month follow-up.

The results of this study will determine whether it is feasible to do a full-scale RCT in the future. If the known beneficial effects of the Managing Fatigue program extend to the PD population, this research will be the evidence needed to support the integration of this novel solution into the care of people with PD.

DETAILED DESCRIPTION:
The aims of this study are to:

Aim 1. Evaluate the feasibility of the IMFP protocol in people living with PD. The sub-aims are to evaluate: (a) the relevance, acceptability, and perceived impact of the content of the MFIP from the perspective of recipients; and (b) the acceptability of the delivery logistics (technology, time, duration) of the MFIP from the perspective of individuals with PD.

Aim 2. Prepare for a full-scale RCT. The sub-aims are to (a) explore the preliminary effectiveness of the MFIP, (b) assess the suitability of the trial recruitment strategy based on the enrolment, completion and attrition rates, and variation in socio-demographic features of participants; (c) evaluate the suitability of potential outcome measures; and (d) use data arising from differences in the study outcomes between the MFIP and control arms to inform a power calculation for the sample size of a definitive RCT. As this study is a feasibility study, there is no primary versus secondary outcomes. The outcomes for this study are occupational performance, occupational balance, fatigue impact, quality of life, sleep quality and self-efficacy.

Sample Size Calculation: As a pilot study, a power calculation is not strictly required. However, in preparation for the current study, investigators conducted both a sample size calculation and consulted previous literature to inform our estimation. To calculate the sample size, the type-1 error was set at 5% and the type-2 error was set at 20% for a power of 80%. Effect sizes were taken from available studies as follows: for the MFI, the effect size of -0.664 and for the COPM the effect size of 0.37. The results indicate that a total sample size of 42 participants will be required using the minimum effect size for the COPM. Estimating an attrition rate of 20%, a convenience sample of 50 participants (25 in each group) will be recruited from across the Halifax Regional Municipality (HRM), Canada.

This sample size selection aligns with recommendations for pilot studies by other researchers who have suggested that a minimum sample size of 24 to 50 is required for pilot feasibility studies. In another study by Hertzog (2008), a minimum sample of 10-25 people per group for feasibility studies is recommended.

Recruitment: Individuals for this study will be recruited in several different ways across the province of Nova Scotia. Investigators will recruit using 1) web-based advertisements on the International Chronic and Complex Conditions Research Group website and KIJIJI, 2) posters at the Parkinson's Society Maritime Region office 3) social media (Twitter, Facebook), 4) public TV advertising and 5) word of mouth. Individuals who are interested in participating in the study will contact the research team.

Individuals who are interested in participating will be invited to contact the research team by email. Potential participants will first undergo an email screening procedure to confirm preliminary eligibility criteria. Once eligibility is confirmed they will be sent study information and a consent form by email. Final eligibility will be confirmed after completion of the FSS and the MMSE during a videoconference call. Consent will be ascertained and confirmed verbally prior to any data collection. Participants will be informed that they may withdraw from the study at any time and for any reason. The assessor for all screening and data collection will be blind to group allocation.

Data Collection-Aim 1: This aim will be achieved using data collected from only the experimental group.

Registered occupational therapists will deliver the IMFP. Therapists graduate with the knowledge and skills to treat people with neurological conditions. All therapists will be required to successfully complete an online training session prior to participation. They will learn about the MFIP and the current evidence-based guidelines and research about working with individuals with PD.

The therapists will be instructed to report to the study supervisor and the principal researcher if there are any safety complications during the sessions.

Feasibility Questionnaires (experimental group only): Two feasibility questionnaires, based on the purposes of the study and the program's intentions, will be administered to participants. Questionnaire # 1 will evaluate the relevance, acceptability, and usability of each session. Participants will complete these, online, after each weekly session. Questionnaire #2 will evaluate the relevance, acceptability, usability, and logistical aspects of the whole program. It will be administered once, at the completion of the program. The responses on the feasibility questionnaires use a five-point Likert scale (Likert, 1932) (0 = 'strongly disagree' to 4 = 'strongly agree). A research assistant, independent from other parts of the study, will send the individualized links for each questionnaire to participants by email. Data collected on the Feasibility Questionnaires will be cleaned and analyzed at the completion of all data collection. This will ensure that this researcher remains masked to group allocation during the study data collection.

Focus Groups: After completion of the program, 15 participants will be recruited to participate in one of three focus groups (n=5) using maximum variation sampling based on disease duration, fatigue severity, and gender. Participants will provide separate consent prior to participating. An experienced, independent research assistant will conduct the focus groups via videoconference using a prepared interview guide. Participants will be encouraged to discuss the feasibility of the program (relevance, usability, acceptability, and logistics), barriers to completion of the program, acceptability of study measures, and any perceived impact/changes (improvements/adverse events).

Data collection - Aim 2: To evaluate the preliminary effectiveness of MFIP in people living with PD and the feasibility of potential outcome measures a collection of patient-reported outcome measures will be used. The outcomes for this study are occupational performance, occupational balance, fatigue impact, quality of life, sleep quality and self-efficacy. Effectiveness data will also be used to inform the power calculation for a definitive trial. The study outcome measures will be administered at baseline, at post-intervention and at three months following completion of the program.

The principal researcher, who will be masked to group allocation, will be responsible for administering all the study outcome measures online using the Opinio Survey Software Application while videoconferencing with the researcher.

Data Analysis: All quantitative data in this study will be analysed using STATA software (release 15 for Windows). After data entry, data will be examined for skewness, outliers, and systematic missing data. Extreme outliers, defined as greater than ±2SD from the mean will be removed from the data if they are less than 5% of all data (Allison, 2001)

Data from the feasibility questionnaires will be analyzed using descriptive analysis, including frequencies and proportions for categorical data (e.g. demographic data), and means, and standard deviations for continuous data (e.g. questionnaires).

Using general linear mixed model analysis, the preliminary effectiveness of the program will be determined. This analysis method will account for missing data at the measurement level. Also, in this study, we do not expect missing data at the item-level as all the measurements are completed with the supervision of the principal researcher. If there are missing data, they will be managed using the required steps based on the protocol of each measurement tool. If the maximum number of missing items has not been included in the protocol of measurements it will be set at 20%. If the scoring algorithm does not provide for missing data, values will be imputed using mean substitution.

Using calculated effect sizes, this study will 1) estimate the preliminary effectiveness and the required sample size for future RCTs, and 2) evaluate the sensitivity and responsiveness of the study outcome measures. Measurement tools with the highest effect size and the smallest significance level are the most sensitive measures to change due to the intervention (Corzillius, Fortin, & Stucki, 1999. In regard to the responsiveness of measures, measurement tools that have higher levels of variability in participants at baseline, in relation to mean change scores, will have a smaller effect and therefore, are less responsive (Husted, Cook, Farewell, & Gladman, 2000. Qualitative data obtained from participants in focus group, together with the quantitative data will be used to recommend outcome measures for the future RCT.

The efficiency of the recruitment strategies will be examined using data from the number of individuals who contact the research team, the number of participants who meet the study criteria, the number who withdraw from the study or are lost to follow-up (attrition rates), and the variation in sociodemographic characteristics of the participants.

Focus groups will be audiotaped and transcribed verbatim. Any potentially identifying information will be removed prior to analysis. Data will be analyzed using the six-stage content analysis framework by Braun and Clarke (2014). Data will be managed using the NVIVO qualitative data analysis software (QSR International Pty Ltd., Version 11, 2015). The text will be coded without any changes in meaning. Coded material will be categorized semantically until themes emerge. Codes and themes will be reviewed and refined until the final distinctive themes can be created (Bob-Milliar, 2014).

ELIGIBILITY:
Inclusion Criteria:

All participants must:

1. Be adults living in Nova Scotia,
2. Self-report Parkinson's disease, and fatigue severe enough to interfere with daily life (measured by a score of ≥4 on the FSS).
3. Read and speak in English
4. Have access to the internet, an electronic device and a private place for Zoom videoconferences.
5. Provide informed consent prior to participation.

Exclusion Criteria:

People will be excluded from the study if :

1. They have previously completed the study program (IMFP )
2. They have co-morbidity that causes severe fatigue (e.g. heart failure, cancer)
3. They indicate a severe cognitive deficit in the MMSE test ( MMSE <13).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Multidimensional Fatigue Inventory (MFI) | Changes from baseline fatigue impact to six weeks later at post-test, and after a three-month follow up.
  Fatigue impact will be measured with the Multidimensional Fatigue Inventory (MFI) (Smets et al., 1995). The MFI is a self-report fatigue tool with 20 items measuring five dimensions: General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motion, and Reduced Activity. Elbers and colleagues (2012) evaluated the MFI in the PD population (N=153). After combining General Fatigue and Physical Fatigue dimensions they reported the reliability and validity of the four-domain scale (Physical Fatigue, Mental Fatigue, Reduced Motivation, and reduced activity) as higher than the original five-domain scale. Testing of the MFI shows good internal consistency (Cronbach's alpha >0.80) and construct validity compared to a Visual Analogue Scale measuring fatigue (0.22<r<0.78) (Smets et al., 1995).
Occupational Balance Questionnaire | Changes from baseline occupational balance to six weeks later, at post-test, and after a three-month follow up.
  Occupational balance will be measured with the Occupational Balance Questionnaire (OBQ) (Wagman & Håkansson, 2014). The OBQ is an 11-item measure developed by Wagman et al., (2014), which assesses individuals' satisfaction and perception with the amount and variation of meaningful occupations. The OBQ measures satisfaction with the amount of time that one takes to accomplish tasks. It uses a 4-level ordinal response scale for each item ranging from 0 "completely disagree" to 3 "completely agree". The OBQ total score ranges from 0 (no occupational balance) to 35 (maximum occupational balance). The psychometric properties of the OBQ have not been explored in PD. However, in the general population, it has shown good internal consistency (Cronbach's alpha= 0.936) and test, re-test reliability (Spearman's Rho= 0.926) for its total score (N=67). Neither ceiling nor floor effects were reported (Håkansson, Wagman, & Hagell, 2019).
Canadian Occupational Performance Measure | Changes from baseline occupational performance to six weeks later, at post-test, and after a three-month follow up.
  Occupational performance will be measured with the Canadian Occupational Performance Measure (COPM) (Law, M. Baptiste, S., Carswell, A. McColl, M. A., Polatajko, H. & Pollock, 1998). The COPM was selected since it has proven to be sensitive to change and was able to detect significant differences between study groups at three months (mean difference =1.2 (95% CI 0.8-1.6) and after 6 months follow-up (mean differences= 0.9 ( 95%CI 0.5-1.3) (I. Sturkenboom et al., 2013). The COPM is a client-centred, standardized, cost-effective, occupation-focused measure used in occupational therapy. It is an individualized outcome measure administered using a semi-structured interview. It measures occupational performance and occupational satisfaction (Law, M. Baptiste, S., Carswell, A. McColl, M. A., Polatajko, H. & Pollock, 1998).
Parkinson's Disease Quality of Life-8 (PDQ-8) | Changes from baseline quality of life to six weeks later, at post-test, and after a three-month follow up.
  Quality of life will be measured with the Parkinson's Disease Quality of Life-8 (PDQ-8) (Tan et al., 2004). The PDQ-8 is a short-form version of the Parkinson Disease Questionaire-39 which assesses the impact of PD on HRQoL over the past month. The PDQ-8 is a summary index with eight items, each representing one dimension of the PDQ-39 (Mobility, Activities of Daily Living, Emotional Well-being, Stigma, Social Support, Cognition, Communication, and Bodily Discomfort). It uses a 0-4 response scale. Scores are summed, then converted into a percentage. Lower scores indicate better quality of life (Peto et al., 1995). The PDQ-8 psychometric properties have been confirmed in several studies (Franchignoni, Giordano, & Ferriero, 2008; Katsarou et al., 2004; Luo et al., 2009; Tan, Luo, Nazri, Li, & Thumboo, 2004). Franchignon et al (2008) and Tan et al (2004) demonstrated good internal consistency (Cronbach's alpha 0.72, 0.81) and construct validity between PDQ-8 and a measure of autonomy and
Pittsburgh Sleep Quality Index (PSQI) | Changes from baseline sleep quality to six weeks later, at post-test, and after a three-month follow up.
  Sleep quality will be measured with the Pittsburgh Sleep Quality Index (PSQI) (Buysse et al., 1989). PSQI is the most common assessment tool used to evaluate sleep quality (Mollayeva et al., 2016). It is a 19-item self-report assessment that measures seven components: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, use of sleep medication, and daytime dysfunction (Buysse, Reynolds, Monk, Berman, & Kupfer, 1989). Component scores range from 0 (no difficulty) to 3 (severe difficulty) and are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality. A meta-analysis by Mollayeva et al. (2016) evaluated the measurement properties of the PSQI. This meta-analysis (N=37) demonstrated that the PSQI has good internal consistency based on Cronbach's alpha, strong reliability and validity, and moderate structural validity in a variety of samples. The PSQI has been used as an outcome measure to test the effectiveness
Self Efficacy for Performing Energy Conservation Strategies Assessment (SEPECSA) | Changes from baseline self-efficacy to six weeks later, at post-test, and after a three-month follow up.
  The Self-efficacy will be measured by the Self Efficacy for Performing Energy Conservation Strategies Assessment (SEPECSA) (Liepold & Mathiowetz, 2005). The SEPECSA was developed based on the Managing Fatigue Program (Liepold & Mathiowetz, 2005) and measures the individual's self-confidence to perform the strategies they learned in the program. The item response scale of the SEPECSA ranges from 1 (not at all confident) to 10 (completely confident). The final score is mean of the item scores. In a study of individuals with MS (N=36), Liepold & Mathiowetz (2005) demonstrated that the SEPECSA has high test and retest reliability (r = .776, ICC = .771), good validity, and very high internal consistency (Cronbach's alpha = .953). The SPECSA has not been used with the PD population, however, it has been used in previous similar studies (Ghahari et al., 2010; Matuska, Mathiowetz, & Finlayson, 2007).

OTHER OUTCOMES:
Relevance, acceptability, and usability of each session of the Individual Managing Fatigue Program | After each weekly session
  The Feasibility Questionnaires 1, developed by the research team based on the purposes of the study and the program's intentions. Feasibility Questionnaire 1 will evaluate the relevance, acceptability, and usability of each session. Participants in the experimental group will complete Feasibility Questionnaire 11 weekly, after each session
Relevance, acceptability, and usability of the Individual Managing Fatigue Program | After six weeks at post test
  The Feasibility Questionnaire 2, developed by the research team, is based on the purposes of the study and the program's intentions. Feasibility Questionnaire #2 will evaluate the relevance, acceptability, usability, and logistical aspects of the whole program at the completion of the program.
Socio-Demographic Questionnaire. | At baseline
  The demographic questionnaire was developed by the research team to inquire about age, gender, living status, current assistive device use, current interventions and medications.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Packer, PhD, Study Director — Dalhousie University
Locations (1):
- Dalhousie University, Halifax, NovaScotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amara AW, Memon AA. Effects of Exercise on Non-motor Symptoms in Parkinson's Disease. Clin Ther. 2018 Jan;40(1):8-15. doi: 10.1016/j.clinthera.2017.11.004. Epub 2017 Dec 1. PMID 29198450
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Beckerman H, Blikman LJ, Heine M, Malekzadeh A, Teunissen CE, Bussmann JB, Kwakkel G, van Meeteren J, de Groot V; TREFAMS-ACE study group. The effectiveness of aerobic training, cognitive behavioural therapy, and energy conservation management in treating MS-related fatigue: the design of the TREFAMS-ACE programme. Trials. 2013 Aug 12;14:250. doi: 10.1186/1745-6215-14-250. PMID 23938046
- [Background] Beiske AG, Svensson E. Fatigue in Parkinson's disease: a short update. Acta Neurol Scand Suppl. 2010;(190):78-81. doi: 10.1111/j.1600-0404.2010.01381.x. PMID 20586741
- [Background] Bivard A, Lillicrap T, Krishnamurthy V, Holliday E, Attia J, Pagram H, Nilsson M, Parsons M, Levi CR. MIDAS (Modafinil in Debilitating Fatigue After Stroke): A Randomized, Double-Blind, Placebo-Controlled, Cross-Over Trial. Stroke. 2017 May;48(5):1293-1298. doi: 10.1161/STROKEAHA.116.016293. Epub 2017 Apr 12. PMID 28404841
- [Background] Blikman LJ, Huisstede BM, Kooijmans H, Stam HJ, Bussmann JB, van Meeteren J. Effectiveness of energy conservation treatment in reducing fatigue in multiple sclerosis: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2013 Jul;94(7):1360-76. doi: 10.1016/j.apmr.2013.01.025. Epub 2013 Feb 8. PMID 23399455
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Chaudhuri A, Behan PO. Fatigue in neurological disorders. Lancet. 2004 Mar 20;363(9413):978-88. doi: 10.1016/S0140-6736(04)15794-2. PMID 15043967
- [Background] Corzillius M, Fortin P, Stucki G. Responsiveness and sensitivity to change of SLE disease activity measures. Lupus. 1999;8(8):655-9. doi: 10.1191/096120399680411416. PMID 10568903
- [Background] Fetters MD, Curry LA, Creswell JW. Achieving integration in mixed methods designs-principles and practices. Health Serv Res. 2013 Dec;48(6 Pt 2):2134-56. doi: 10.1111/1475-6773.12117. Epub 2013 Oct 23. PMID 24279835
- [Background] Cup EH, Scholte op Reimer WJ, Thijssen MC, van Kuyk-Minis MA. Reliability and validity of the Canadian Occupational Performance Measure in stroke patients. Clin Rehabil. 2003 Jul;17(4):402-9. doi: 10.1191/0269215503cr635oa. PMID 12785249
- [Background] Dedding C, Cardol M, Eyssen IC, Dekker J, Beelen A. Validity of the Canadian Occupational Performance Measure: a client-centred outcome measurement. Clin Rehabil. 2004 Sep;18(6):660-7. doi: 10.1191/0269215504cr746oa. PMID 15473118
- [Background] DeLuca J, Genova HM, Capili EJ, Wylie GR. Functional neuroimaging of fatigue. Phys Med Rehabil Clin N Am. 2009 May;20(2):325-37. doi: 10.1016/j.pmr.2008.12.007. PMID 19389614
- [Background] Elbers RG, Berendse HW, Kwakkel G. Treatment of Fatigue in Parkinson Disease. JAMA. 2016 Jun 7;315(21):2340-1. doi: 10.1001/jama.2016.5260. PMID 27272586
- [Background] Elbers RG, van Wegen EE, Verhoef J, Kwakkel G. Reliability and structural validity of the Multidimensional Fatigue Inventory (MFI) in patients with idiopathic Parkinson's disease. Parkinsonism Relat Disord. 2012 Jun;18(5):532-6. doi: 10.1016/j.parkreldis.2012.01.024. Epub 2012 Feb 22. PMID 22361576
- [Background] Elbers RG, van Wegen EE, Verhoef J, Kwakkel G. Impact of fatigue on health-related quality of life in patients with Parkinson's disease: a prospective study. Clin Rehabil. 2014 Mar;28(3):300-11. doi: 10.1177/0269215513503355. Epub 2013 Oct 10. PMID 24113725
- [Background] Eyssen IC, Beelen A, Dedding C, Cardol M, Dekker J. The reproducibility of the Canadian Occupational Performance Measure. Clin Rehabil. 2005 Dec;19(8):888-94. doi: 10.1191/0269215505cr883oa. PMID 16323388
- [Background] Finlayson M, Preissner K, Cho C, Plow M. Randomized trial of a teleconference-delivered fatigue management program for people with multiple sclerosis. Mult Scler. 2011 Sep;17(9):1130-40. doi: 10.1177/1352458511404272. Epub 2011 May 11. PMID 21561960
- [Background] Foster ER, Golden L, Duncan RP, Earhart GM. Community-based Argentine tango dance program is associated with increased activity participation among individuals with Parkinson's disease. Arch Phys Med Rehabil. 2013 Feb;94(2):240-9. doi: 10.1016/j.apmr.2012.07.028. Epub 2012 Aug 15. PMID 22902795
- [Background] Franchignoni F, Giordano A, Ferriero G. Rasch analysis of the short form 8-item Parkinson's Disease Questionnaire (PDQ-8). Qual Life Res. 2008 May;17(4):541-8. doi: 10.1007/s11136-008-9341-6. PMID 18415705
- [Background] Franssen M, Winward C, Collett J, Wade D, Dawes H. Interventions for fatigue in Parkinson's disease: A systematic review and meta-analysis. Mov Disord. 2014 Nov;29(13):1675-8. doi: 10.1002/mds.26030. Epub 2014 Sep 18. PMID 25234443
- [Background] Friedman JH, Abrantes A, Sweet LH. Fatigue in Parkinson's disease. Expert Opin Pharmacother. 2011 Sep;12(13):1999-2007. doi: 10.1517/14656566.2011.587120. Epub 2011 Jun 3. PMID 21635199
- [Background] Friedman JH, Brown RG, Comella C, Garber CE, Krupp LB, Lou JS, Marsh L, Nail L, Shulman L, Taylor CB; Working Group on Fatigue in Parkinson's Disease. Fatigue in Parkinson's disease: a review. Mov Disord. 2007 Feb 15;22(3):297-308. doi: 10.1002/mds.21240. PMID 17133511
- [Background] Friedman JH. Fatigue in Parkinson's disease patients. Curr Treat Options Neurol. 2009 May;11(3):186-90. doi: 10.1007/s11940-009-0022-8. PMID 19364453
- [Background] Ghahari S, Packer TL, Passmore AE. Development, standardisation and pilot testing of an online fatigue self-management program. Disabil Rehabil. 2009;31(21):1762-72. doi: 10.1080/09638280902751956. PMID 19479510
- [Background] Ghahari S, Leigh Packer T, Passmore AE. Effectiveness of an online fatigue self-management programme for people with chronic neurological conditions: a randomized controlled trial. Clin Rehabil. 2010 Aug;24(8):727-44. doi: 10.1177/0269215509360648. Epub 2010 Jun 11. PMID 20543022
- [Background] Golab-Janowska M, Kotlega D, Safranow K, Meller A, Budzianowska A, Honczarenko K. Risk Factors of Fatigue in Idiopathic Parkinson's Disease in a Polish Population. Parkinsons Dis. 2016;2016:2835945. doi: 10.1155/2016/2835945. Epub 2016 Jan 26. PMID 26925292
- [Background] Goodwin VA, Richards SH, Taylor RS, Taylor AH, Campbell JL. The effectiveness of exercise interventions for people with Parkinson's disease: a systematic review and meta-analysis. Mov Disord. 2008 Apr 15;23(5):631-40. doi: 10.1002/mds.21922. PMID 18181210
- [Background] Hakansson C, Wagman P, Hagell P. Construct validity of a revised version of the Occupational Balance Questionnaire. Scand J Occup Ther. 2020 Aug;27(6):441-449. doi: 10.1080/11038128.2019.1660801. Epub 2019 Sep 14. PMID 31524026
- [Background] Havlikova E, Rosenberger J, Nagyova I, Middel B, Dubayova T, Gdovinova Z, van Dijk JP, Groothoff JW. Impact of fatigue on quality of life in patients with Parkinson's disease. Eur J Neurol. 2008 May;15(5):475-80. doi: 10.1111/j.1468-1331.2008.02103.x. Epub 2008 Mar 5. PMID 18325024
- [Background] Herlofson K, Larsen JP. The influence of fatigue on health-related quality of life in patients with Parkinson's disease. Acta Neurol Scand. 2003 Jan;107(1):1-6. doi: 10.1034/j.1600-0404.2003.02033.x. PMID 12542506
- [Background] Hugos CL, Copperman LF, Fuller BE, Yadav V, Lovera J, Bourdette DN. Clinical trial of a formal group fatigue program in multiple sclerosis. Mult Scler. 2010 Jun;16(6):724-32. doi: 10.1177/1352458510364536. Epub 2010 Apr 7. PMID 20375125
- [Background] Katsarou Z, Bostantjopoulou S, Peto V, Kafantari A, Apostolidou E, Peitsidou E. Assessing quality of life in Parkinson's disease: can a short-form questionnaire be useful? Mov Disord. 2004 Mar;19(3):308-12. doi: 10.1002/mds.10678. PMID 15022185
- [Background] Kluger BM. Fatigue in Parkinson's Disease. Int Rev Neurobiol. 2017;133:743-768. doi: 10.1016/bs.irn.2017.05.007. Epub 2017 Jun 20. PMID 28802940
- [Background] Kos D, Duportail M, D'hooghe M, Nagels G, Kerckhofs E. Multidisciplinary fatigue management programme in multiple sclerosis: a randomized clinical trial. Mult Scler. 2007 Sep;13(8):996-1003. doi: 10.1177/1352458507078392. Epub 2007 Jul 10. PMID 17623738
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Zesiewicz TA, Patel-Larson A, Hauser RA, Sullivan KL. Social Security Disability Insurance (SSDI) in Parkinson's disease. Disabil Rehabil. 2007 Dec 30;29(24):1934-6. doi: 10.1080/09638280701257247. Epub 2007 Jul 3. PMID 17852221
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Wagman P, Hakansson C. Introducing the Occupational Balance Questionnaire (OBQ). Scand J Occup Ther. 2014 May;21(3):227-31. doi: 10.3109/11038128.2014.900571. Epub 2014 Mar 21. PMID 24649971
- [Background] Vanage SM, Gilbertson KK, Mathiowetz V. Effects of an energy conservation course on fatigue impact for persons with progressive multiple sclerosis. Am J Occup Ther. 2003 May-Jun;57(3):315-23. doi: 10.5014/ajot.57.3.315. PMID 12785670
- [Background] Van Heest KNL, Mogush AR, Mathiowetz VG. Effects of a One-to-One Fatigue Management Course for People With Chronic Conditions and Fatigue. Am J Occup Ther. 2017 Jul/Aug;71(4):7104100020p1-7104100020p9. doi: 10.5014/ajot.2017.023440. PMID 28661378
- [Background] van den Akker LE, Beckerman H, Collette EH, Eijssen IC, Dekker J, de Groot V. Effectiveness of cognitive behavioral therapy for the treatment of fatigue in patients with multiple sclerosis: A systematic review and meta-analysis. J Psychosom Res. 2016 Nov;90:33-42. doi: 10.1016/j.jpsychores.2016.09.002. Epub 2016 Sep 7. PMID 27772557
- [Background] Packer TL, Brink N, Sauriol A. Managing Fatigue: A six-week course for energy conservation. Therapy Skill Builders: Tucson, Ariz. 1995
- [Derived] Alizadeh N, Packer TL, Jaswal S, Sturkenboom I, Warner G. Client Perceptions of the Individual Packer Managing Fatigue Program: A Mixed-Method Evaluation. OTJR (Thorofare N J). 2024 Oct;44(4):632-641. doi: 10.1177/15394492241262740. Epub 2024 Jul 31. PMID 39086144

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT04267107/Prot_SAP_001.pdf
  • Informed Consent Form (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT04267107/ICF_000.pdf